CLINICAL TRIAL: NCT05255731
Title: Effect of the Low Power Laser in the Treatment of Pain After the Third Molar Lower Extraction. A Randomised Single-blind Clinical Trial Split-mouth
Brief Title: Effect of Low Power Laser in the Pain After Lower Tooth Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Mario Pérez Sayáns, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCT-PBM/TM-USC/UB-22
Record Dates: First submitted 2022-02-01; First posted 2022-02-24 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Third Molar Extraction; Oral Pain; Tooth Extraction
Keywords: Dentistry; Tooth extraction; Photobiomodulation; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: One side the laser off will be applied, on the other side, the laser on will be applied,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Group (GL) (Active Comparator): Patients will be submitted to a low power laser application immediately after suturing of the surgical area. The radiation emission shall be conducted according to protocol.
  Interventions: Radiation: Low frequency laser activated photobiomodulation
- Control Group (CG) (Placebo Comparator): In these patients the investigators will use the same protocol applied in the experimental group (time and application values) but the laser device will be turn off.
  Interventions: Other: Low frequency laser photobiomodulation inactive

INTERVENTIONS:
Radiation: Low frequency laser activated photobiomodulation — Protocol description Infrared: analgesia, biostimulation of tissues, edema and hyperemia (hard and soft tissues). There will be 11 laser application points, 3 intra-oral and 8 extra-oral, with a total dose of 33J.
  Intraoral: one point in the region of the mandibular lingula (point of submersion of the mandibular nerve), one vestibular point and one lingual point in relation to the alveolus of the extracted wisdom tooth.
  Extraoral: for muscle relaxation, five points on the masseter muscle; for oedema drainage, one point in each lymph node region: parotid, submandibular and buccal.
  Arms: Laser Group (GL)
Other: Low frequency laser photobiomodulation inactive — The same protocol as the activated group
  Arms: Control Group (CG)

SUMMARY:
Introduction: Previously published studies report a prevalence ranging from 35.9% to 58.7% of the general population with at least one impacted wisdom tooth. Surgical extraction of wisdom teeth is the procedure most often associated with postoperative complications, such as pain, swelling, trismus, and oral discomfort during the first postoperative days. These complications arise from an inflammatory response, which is a direct and immediate consequence of the surgical intervention and can limit the patients' daily functions in the recovery phase and compromise their quality of life. Several methods have been used to control postoperative morbidity related to wisdom tooth extraction, including administration of proteolytic enzymes, tube drains, cryotherapy, anti-inflammatory and analgesic drugs and low level laser therapy.

Objectives: To test whether the use of low power laser can improve post-operative pain, swelling and healing of the surgical wound.

Material and methods: A double-centre, randomised, split-mouth, double-centre clinical study will be carried out in 38 patients per centre, totalling 76 patients and 152 wisdom teeth, who will undergo surgery for the extraction of the lower third molars. The necessary data for the study will be taken on the days of the consultation for surgery planning, on the day of surgery, by the patient on each post-operative day and on the 7th post-operative day (at the time of suture removal ).

ELIGIBILITY:
Inclusion Criteria:

* Patients who require extraction of the two lower wisdom teeth due to previous infection or pain, orthodontics or crowding, caries and who have a similar degree of difficulty according to the Pell and Gregory/Winter classifications.
* Patients must have the capacity to understand and decide at the time of voluntarily signing the informed consent before any intervention related to the study is performed.
* Patients who, after being informed about the aims and procedures of the research, agree and sign the informed consent form. Patients must be willing and able to adhere to the study in order to complete the necessary visits.

Exclusion Criteria:

* Patients with uncontrolled systemic disease (ASA ≥ III).
* Patients with severe periodontal disease or acute pericoronitis.
* Smokers of more than 5 cigarettes per day.
* Pregnant and lactating women, as the effect of laser therapy in this population has not been studied, its use is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluate edema after surgery | 7 days
  To evaluate the effect of diode laser radiation of 808 nm (infrared) applied intra and extra-orally on the post-operative edema (by measuring in centimetres obtained by a ruler - external contour of the face from the tragus to the labial comisure, from the gonion to the external ocular corner, the greater the measurement obtained, when compared with the initial measurement, the greater the post-operative edema).

SECONDARY OUTCOMES:
Reported pain | 7 days
  The degree of pain reported by patients using a visual analogue scale (VAS). Scale from 0 to 10, where zero means no pain and ten means severe pain
Rescue medication for pain | 7 days
  To assess whether there has been a change in the amount of pills consumed as rescue medication for pain management. Through the number of pills used by the patient after each surgery.
Trismus | 7 days
  With a ruler the distance of the maximum opening between the upper right and lower right central incisors before surgery will be measured (the measurement in centimetres). The smaller the measurement of mouth opening obtained, compared to the initial measurement, the greater the post-operative trismus)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will anonymize and categorize the clinical data of the patients to share the information with the other researchers of the group.